CLINICAL TRIAL: NCT05679024
Title: Stroke Prophylaxis With Apixaban in Chronic Kidney Disease Stage 5 Patients With Atrial Fibrillation
Acronym: SACK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU CT 2022-501600-10-00
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Diseases; Atrial Fibrillation; Stroke; Intracerebral Hemorrhage; Major Bleed; Cardiovascular Complication; Death; Kidney Transplant; Complications; Thromboses, Venous
Keywords: Chronic kidney disease; Hemodialysis; Peritoneal dialysis; Kidney transplantation; Atrial fibrillation; Oral anticoagulation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Atrial Fibrillation; Stroke; Cerebral Hemorrhage; Death; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Pragmatic Prospective Open Label Parallel-Group Multicenter Phase 3b Randomized Controlled Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apixaban 2.5 mg twice daily and standard of care (Active Comparator): Apixaban 2.5 mg twice daily (low dose) and all other standard of care
  Interventions: Drug: Apixaban 2.5 milligram Oral Tablet
- Standard of care and no anticoagulation (No Intervention): All other Standard of care and no anticoagulation

INTERVENTIONS:
Drug: Apixaban 2.5 milligram Oral Tablet — Oral Tablet
  Arms: Apixaban 2.5 mg twice daily and standard of care

SUMMARY:
Objective: To study the efficacy and safety of apixaban as stroke prophylaxis in patients with chronic kidney disease (CKD) stage 5 and atrial fibrillation (AF) with or without dialysis treatment. The study hypothesis is that compared to no anticoagulation, apixaban reduces the incidence of ischemic stroke without causing an unacceptable increase in fatal or intracranial bleeding events.

The secondary objectives are to evaluate the risk of all-cause mortality, cardiovascular events, and major bleeding in people with CKD stage 5 and AF treated with apixaban compared to standard of care without anticoagulation.

Trial design: Pragmatic Prospective Open Label Randomized Controlled Clinical Trial, phase 3b over 12-72 months.

Trial population: 1000-1400 patients at ≈50 sites in Sweden, Finland, Norway, Iceland and Poland Eligibility criteria: Adults ≥18 years with CKD stage 5 (ongoing treatment with any chronic dialysis treatment OR an estimated glomerular filtration rate (eGFR)* <20 ml/min/1.73 m2 at least twice 3 months apart of which at least one occasion is <15 ml/min/1.73 m2 due to CKD during the last 12 months) and a diagnosis of chronic, paroxysmal, persistent, or permanent AF or atrial flutter (AFL) with CHA2DS2-VASc score ≥2 for men or ≥3 or more for women as an indication for oral anticoagulation.

The exclusion criteria are AF or AFL due to reversible causes, rheumatic mitral stenosis or moderate-to-severe non-rheumatic mitral stenosis at the time of inclusion into the study, a condition other than AF or AFL that requires chronic anticoagulation, contraindications for anticoagulation, active bleeding or serious bleeding within 3 months, planned for surgery within 3 months, and current use of strong inhibitors of both CYP3A4 and P-glycoprotein.

Interventions: Randomization 1:1 to treatment with apixaban 2.5 mg twice daily and standard of care, or standard of care and no anticoagulation.

Outcome measures: primary efficacy (time to first ischemic stroke); primary safety (the composite of time to first intracranial bleeding or fatal bleeding); secondary efficacy (time to all-cause mortality, time to cardiovascular event or cardiovascular death); secondary safety (time to first major bleeding according to International Society on Thrombosis and Hemostasis (ISTH) criteria)

DETAILED DESCRIPTION:
Background and rationale: Atrial fibrillation (AF) is common (15-30%) in patients with chronic kidney disease (CKD) and AF prevalence increases with severity of CKD. In late stages of CKD, randomized control trials (RCT) of both efficacy and safety of any anticoagulation therapy, both warfarin and direct oral anticoagulation (DOAC) drugs, for stroke prophylaxis in AF are lacking. The efficacy of warfarin and DOACs have been evaluated in observational trials in patients with stage 5 CKD, but the results have been conflicting, and these studies were all subjected to selection bias in one way or the other. Instead, observational studies have demonstrated several adverse side-effects. Among them an increased number of bleedings including hemorrhagic stroke in patients treated with warfarin, and calciphylaxis, a very serious complications unknown in the normal population linked to the withdrawal of vitamin-K-dependent protection of vascular calcification in CKD. With apixaban treatment several benefits were reported. Firstly, a potential protective effect against ischemic stroke. Secondly, a lower incidence of bleeding complications as observed in the major trials, and thirdly, no disturbance in vitamin K turnover as compared to warfarin treatment. In addition, apixaban treatment does not require routine monitoring and have fewer drug/food interactions. For patients with CKD stage 5, treatment with apixaban appears to have a lower bleeding risk than warfarin treatment.

Rationale to study design: There are no previous randomized controlled clinical trials in this study population. The SACK study is conducted in approximately 50 sites in Sweden, Finland, Norway, Iceland and Poland, and additional European countries, if necessary. In Sweden, the study will be register-randomized (via the national Swedish Renal Register [SNR]) whereas the other countries in the study will include patients in a traditional way for clinical trials.

The study design will be an individually randomized two-armed parallel-group design. Apixaban will be prescribed and renewed by the local investigator via regular prescription or distributed by the investigating site at regular intervals in all participating countries. Due to open-label prescription and safety reasons, the study will be conducted as an open-label trial with end-point evaluation. Patients who are randomized to apixaban and those who are randomized to standard of care with no anti-coagulation will receive all other guideline-recommended standard of care treatments. Patients already on prior warfarin or apixaban therapy, or on regular low molecular weight heparin (LMWH) can also be randomized to either treatment arm (their current anticoagulation is discontinued at the inclusion visit) after an individualized risk assessment. At inclusion, patients will provide routine blood samples including hemoglobin, eGFR, and coagulation parameters.

The end of the clinical study for each individual patient is defined as the End of Study (EoS) visit. The EoS for a patient is after 72 months or when 247 primary events have been reached, whichever comes first. An interim analysis will take place after 1000 patient-years with the purpose to evaluate event rate and to be able to closer determine the exact number of patients and duration of the trial. The end of the clinical trial is defined as the last visit of the last subject in the study (LVLS).

A Data and Safety Monitoring Board (DSMB) will supervise this study, and primary safety and efficacy endpoints and major bleedings will additionally be evaluated by independent external reviewers according to a predefined Central Event Adjudication charter.

Exploratory outcomes: Time to first thromboembolic event defined as a composite of deep vein thrombosis, pulmonary embolism, transient ischemic attack Time to dialysis access thrombosis Time to kidney replacement therapy Delayed graft function in patients undergoing kidney transplantation Thrombosis of renal artery or vein in patients undergoing kidney transplantation

Among the secondary safety outcomes are time to major bleeding according to ISTH criteria. We are especially interested in the safety outcomes of the subgroup undergoing a kidney transplantation from the waiting list and therefore we have an extended protocol for those participants.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. 18 years of age or older
3. Ongoing treatment with any chronic dialysis treatment OR an estimated glomerular filtration rate (eGFR)* <20 ml/min/1.73 m2 at least twice 3 months apart of which at least one occasion is <15 ml/min/1.73 m2 due to CKD during the last year (12 months).
4. Diagnosis of chronic (i.e., repeated) paroxysmal, persistent, or permanent atrial fibrillation (AF) or atrial flutter (AFL)
5. CHA2DS2-VASc score ≥2 or more for men ≥3 or more for women as an indication for oral anticoagulation
6. Women of childbearing potential (WOCBP) should have a negative highly effective pregnancy test at screening and must agree to follow instructions for method(s) of contraception for the duration of treatment

Exclusion Criteria:

Participants may not be included in the study if any of the following criteria are met:

1. AF or AFL due to reversible causes (e.g., thyrotoxicosis, pericarditis)
2. Any degree of rheumatic mitral stenosis or moderate-to-severe non-rheumatic mitral stenosis at the time of inclusion into the study
3. Any condition other than AF or AFL that requires chronic anticoagulation (e.g., a prosthetic mechanical heart valve, antiphospholipid syndrome).
4. Any contraindication for anticoagulation including

   1. endocarditis
   2. documented intolerance for apixaban
   3. liver disease with documented coagulation disorder
   4. pregnancy or breast feeding
5. Active bleeding or serious bleeding within 3 months, or

   1. documented hemorrhagic blood dyscrasia
   2. patients currently receiving dual antiplatelet therapy
6. Planned for surgery

   1. kidney transplantation with a living donor within 3 months
   2. active on the kidney transplant waiting list at a kidney transplant center where apixaban use is prohibited
   3. valvular heart disease surgery
7. Current use of strong inhibitors of both CYP3A4 and P-glycoprotein in accordance with the summary of product characteristics (SmPC) of apixaban or regular intake of non-steroidal anti-inflammatory drugs (NSAID) or cyclooxygenase-2 (COX2) inhibitors
8. Any condition or circumstance in which the patient should not participate in the study according to the study investigator (reason documented in the pre-screening protocol)

Being active on the kidney transplant waiting list is not an exclusion criterion if it is allowed according to the current clinical guidelines at the transplant clinic where the patient is registered. The patient must report changes in waiting list status to the investigator promptly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke or systemic embolism (efficacy) | Up to 72 months
  Time to ischemic stroke or systemic embolism
Intracranial bleeding (including hemorrhagic stroke) and fatal bleeding (safety) | Up to 72 months
  Time to intracranial or fatal bleeding

SECONDARY OUTCOMES:
All-cause mortality | Up to 72 months
  Time to death
Cardiovascular event | Up to 72 months
  Composite of time to myocardial infarction, cardiovascular intervention or cardiovascular death
Individual components of cardiovascular event | Up to 72 months
  Time to myocardial infarction and cardiovascular intervention and cardiovascular death
Major bleeding | Up to 72 months
  Time to major bleeding according to ISTH criteria (modified)
Major bleeding in patients undergoing kidney transplantation | Up to 72 months
  Time to major surgical bleeding according to ISTH criteria

OTHER OUTCOMES:
Thromboembolic event | Up to 72 months
  Time to transitory ischemic attack, pulmonary embolism, deep vein thrombosis,
Dialysis access thrombosis | Up to 72 months
  Time to dialysis access thrombosis
Kidney replacement therapy initiation | Up to 72 months
  Time to Kidney replacement therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Marie Evans, Ass Prof, Principal Investigator — Karolinska University Hospital; Maria Svensson, Prof, Study Chair — Uppsala University
Locations (34):
- Finland (3):
  - Helsingfors University hospital, Helsinki
  - Tampere hospital, Tampere
  - Turku hospital, Turku
- Landspitali, the National University hospital of Iceland, Reykjavik, Iceland
- Norway (5):
  - Oslo Akershus, Oslo
  - Oslo Universitetssjukhus Ullevål, Oslo
  - Stavanger hospital, Stavanger
  - Tromsö hospital, Tromsø
  - Vestfold hospital, Tønsberg
- Sweden (25):
  - Falun hospital, Falun, Dalarna County
  - Östersund hospital, Östersund, Jämtland County
  - Lasarettet i Falun, Falun, Region Dalarna
  - Mora sjukhus, Mora, Region Dalarna
  - Länssjukhuset Kalmar, Kalmar, Region Kalmar Län
  - Kalix hospital, Kalix, Region Norrbotten
  - Skånes University hospital Lund, Lund, Region Skåne
  - Skånes University hospital Malmö, Malmo, Region Skåne
  - Norrland University hospital Umeå, Umeå, Region Västerbotten
  - Sundsvall, Sundsvall, Region Västernorrland
  - Västmanlands sjukhus Västerås, Västerås, Region Västmanland
  - Borås sjukhus, Borås, Region Västra Götaland
  - Sahlgrenska University hospital, Gothenburg, Region Västra Götaland
  - Skaraborg hospital Skövde, Skövde, Region Västra Götaland
  - University hospital Örebro, Örebro, Region Örebro Län
  - Linköping University hospital, Linköping, Region Östergötland
  - Länssjukhuset Ryhov, Jönköping
  - Karlshamns sjukhus, Karlshamn
  - Karlstad Central hospital, Karlstad
  - Norrköpings sjukhus, Norrköping
  - Skellefteå hospital, Skellefteå
  - Karolinska Universitetssjukhuset, Stockholm
  - Danderyd sjukhus AB, Stockholm
  - Akdemiska sjukhuset Uppsala, Uppsala
  - Varberg hospital, Varberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593